CLINICAL TRIAL: NCT06343389
Title: Study of Acute Kidney Injury in Patients With Liver Cirrhosis at Sohag University Hospital
Brief Title: Acute Kidney Injury in Patients With Liver Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Shehab Ahmed, Sohag, Egypt, Sohag University
Other Study IDs: Soh-Med-24-03-14MS
Record Dates: First submitted 2024-03-25; First posted 2024-04-02 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury in Patients With Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: Cirrhotic patients with Acute kidney injury
  Interventions: Diagnostic Test: serum creatinine
- group B: Cirrhotic patients without Acute kidney injury
  Interventions: Diagnostic Test: serum creatinine

INTERVENTIONS:
Diagnostic Test: serum creatinine — to detect patients with Acute kidney injury

SUMMARY:
In our locality, limited studies have discussed AKI in patients with liver cirrhosis and its outcome, therefore we aim to highlight the incidence, patterns, risk factors, and outcomes of acute kidney injury in patients with liver cirrhosis at Sohag University Hospital.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common condition in patients with cirrhosis. It occurs in up to 50% of hospitalized patients with cirrhosis and in 58% of such patients in the intensive care unit. AKI is one of the key predictors for short-term mortality in patients with liver cirrhosis with mortality rates as high as 90%. There is a remarkable increase in length of hospital stay with high financial burden on patients with AKI.

In general, the three main causes of AKI are renal hypoperfusion (also referred to as prerenal AKI), which in most cases is due to hypovolemia; intrinsic, structural kidney injury; and postrenal injury due to urinary obstruction. A unique cause of AKI due to renal hypoperfusion in patients with cirrhosis is the hepatorenal syndrome (HRS), which is the result of renal vasoconstriction. Early identification and management of AKI may improve outcomes.

In our locality, limited studies have discussed AKI in patients with liver cirrhosis and its outcome, therefore we aim to highlight the incidence, patterns, risk factors, and outcomes of acute kidney injury in patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients ( age more than 18 years old ) in Sohag University Hospital

Exclusion Criteria:

* patients with known preexisting chronic kidney disease
* patients who had undergone renal transplantation
* malignancy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients ( age more than 18 years old ) in Sohag University Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury in cirrhotic patients in Sohag University Hospital | 1 year
  Number of new cases of acute kidney injury (which will be diagnosed by either increase in serum creatinine ≥0.3 mg/dl within 48 hours; or, a percentage increase in serum creatinine ≥50% within the prior seven days) occurring in cirrhotic patients in Sohag University Hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt